CLINICAL TRIAL: NCT04205461
Title: Prospective Evaluation of Programmed Ventricular Stimulation Before Pulmonary Valve Replacement in Patients With Tetralogy of Fallot
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Paris Cardiovascular Research Center (Inserm U970) (Other Government)
Collaborators: European Georges Pompidou Hospital (Other); Centre Chirurgical Marie Lannelongue (Other); Clinique Pasteur Toulouse (Other); Hopital Louis Pradel (Other); Hôpital Necker-Enfants Malades (Other)
Responsible Party: Sponsor
Other Study IDs: ParisCardioRC
Record Dates: First submitted 2019-12-15; First posted 2019-12-19 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Congenital Heart Disease; Fallot Tetralogy; Ventricular Arrythmia; Pulmonary Valve Regurgitation
Keywords: programmed ventricular stimulation; catheter ablation; electrophysiology study; tetralogy of Fallot; pulmonary valve replacement
MeSH Terms: conditions — Heart Defects, Congenital; Tetralogy of Fallot; Pulmonary Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Programmed ventricular stimulation before PVR
  Interventions: Procedure: Programmed ventricular stimulation

INTERVENTIONS:
Procedure: Programmed ventricular stimulation — Programmed ventricular stimulation before pulmonary valve replacement. Voltage and activation mapping of right ventricle in a subset of patients.

SUMMARY:
Severe pulmonary regurgitation is common in patients with Tetralogy of Fallot and results in progressive right ventricular dilatation and dysfunction. Pulmonary valve replacement is frequent in this population, and percutaneous procedures are increasing.

Ventricular arrhythmias are a frequent late complication in patients with tetralogy of Fallot. The most common critical isthmus of ventricular tachycardias is between the pulmonary valve and the ventricular septal defect patch.

While an electrophysiology study is sometimes performed in expert centers before surgical pulmonary valve replacement to guide a surgical ablation if needed, this approach is not recommended in current guidelines. An electrophysiology study should also be considered before percutaneous pulmonary valve replacement, as a part of the critical isthmus may be covered by the prosthetic pulmonary valve. Moreover, ablation after percutaneous pulmonary valve insertion exposes patients to the risks of traumatic valve or stent injury and infectious endocarditis.

At present, reliable predictors to identify high-risk patients in whom an electrophysiology study should be performed before pulmonary valve replacement are lacking.

The aim of this study is to assess prospectively the yield of systematic electrophysiology study and programmed ventricular stimulation before surgical and percutaneous pulmonary valve replacement in patients with tetralogy of Fallot.

ELIGIBILITY:
Inclusion Criteria:

* All patients with repaired tetralogy of Fallot referred for surgical or percutaneous pulmonary valve replacement

Exclusion Criteria:

* Absence of patient's consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with repaired tetralogy of Fallot referred for surgical or percutaneous pulmonary valve replacement
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive programmed ventricular stimulation defined as inducibility of sustained ventricular tachycardia or fibrillation | During ventricular programmed stimulation
  Rate of sustained monomorphic or polymorphic ventricular tachycardia or ventricular fibrillation sustained > 30 secondes during programmed ventricular stimulation

SECONDARY OUTCOMES:
Critical isthmus involved in ventricular tachycardias induced | During ventricular programmed stimulation
  Description of different critical isthmus involved in ventricular tachycardias induced. Electrophysiological characteristics will be analyzed (conduction velocity, voltage, fragmentation, lenght, width).
Complications associated with programmed ventricular stimulation | 1 month
  Complications considered:
  * death
  * vascular complications
  * pericardial effusion
  * stroke
  * atrioventricular block
  * heart failure
Rate of ventricular arrhythmias during the follow-up after pulmonary valve replacement | 24 months
  Sustained ventricular tachycardias or ventricular fibrillations > 30 secondes and sudden cardiac deaths will be considered

CONTACTS AND LOCATIONS:
Overall Officials: Victor Waldmann, MD, MPH, Principal Investigator — European Georges Pompidou Hospital
Locations (1):
- Paris Cardiovascular Research Center, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Waldmann V, Bessiere F, Gardey K, Bakloul M, Belli E, Bonnet D, Chaussade AS, Cohen S, Delasnerie H, Dib N, Di Filippo S, Dulac A, Hascoet S, Henaine R, Iserin L, Karsenty C, Ladouceur M, Legendre A, Malekzadeh-Milani S, Mostefa Kara M, Radojevic J, Ratsimandresy M, Marijon E, Maltret A, Khairy P, Combes N. Systematic Electrophysiological Study Prior to Pulmonary Valve Replacement in Tetralogy of Fallot: A Prospective Multicenter Study. Circ Arrhythm Electrophysiol. 2023 Jun;16(6):e011745. doi: 10.1161/CIRCEP.122.011745. Epub 2023 May 12. PMID 37170812